CLINICAL TRIAL: NCT06572332
Title: Simulation-informed Modelling and Personalized Evaluation (SIMPLE): A Computational Study of MRI-based Brain Age Matrices
Brief Title: Simulation-informed Modelling and Personalized Evaluation (SIMPLE) in Ageing Populations
Status: Enrolling by invitation | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, LU Hanna, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2023.171
Record Dates: First submitted 2024-08-25; First posted 2024-08-27 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Neurodegenerative Diseases; Aging; Brain; Cognitive Dysfunction
Keywords: MRI; Brain age; Deep learning; Healthy longevity; Resilence; Cognitive maintenance; Simulation; Imaging phenotypes
MeSH Terms: conditions — Neurodegenerative Diseases; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multimodal magnetic resonance imaging (MRI), detecting brain structural and functional changes, has emerged as a powerful and promising technique to study individual's brain, as T1-weighted scans can detect morphometric features, diffusion tensor imaging (DTI) scans can quantify structural connectivity, and functional MRI can capture the features of functional connectivity. Notably, with the advances in quantitative methods, computational models of brain age and brain-predicted age difference (brain-PAD) detecting the ageing effects on individual's brain features are becoming increasingly popular in clinical studies, which might revolutionize the diagnostic and prognostic phonotypes of age-related brain diseases globally.

DETAILED DESCRIPTION:
The score of brain-PAD has threefold explanations: a. negative score representing decelerated brain ageing (brain age<chronological age); b. positive score representing accelerated brain ageing (brain age>chronological age); c. score equal to zero, representing normal brain ageing (brain age=chronological age). The score of brain-PAD indicates the brain ageing pattern with the interaction of lifestyle and cognitive status at individual level. For example, based on structural MRI scans, a younger brain age or a negative score of brain-PAD was found to be associated with better cognition, which indicates the potential utilities of brain age matrices in predicting individual's cognitive maintenance and healthy longevity

ELIGIBILITY:
Inclusion Criteria:

* Chinese old adults are the ones who are over 60 years of chronological age.
* Sleep disturbance: individual's subjective sleep quality is assessed using the Pittsburgh Sleep Quality Index (PSQI) with a total score >5.

Exclusion Criteria:

* History of bipolar disorders or psychosis.
* History of major neurological deﬁcits, including stroke, transient ischemic attack or brain tumor.
* Unable to participant magnetic resonance imaging (MRI) scanning.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ageing adults and adults with sleep disturbances.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Estimated brain age | Baseline
  Using the structural and functional connectivity, individual's brain age is calculated based on the connectivity features of core brain networks.
Cognitive maintenance | Baseline
  The dynamic change of cognitive status is used to evaluate cognitive maintenance. The performance of global cognition is used to determine the cognitive status, including mild neurocognitive disorder (NCD) and major NCD. The global cognition is measured by mini-mental state examination (MMSE).
Plasma β-amyloid | Baseline
  The levels of Aβ42 and Aβ40 in the plasma samples will be quantified by enzyme-linked immunosorbent assay.

SECONDARY OUTCOMES:
Brain-predicted age difference (brain-PAD) | Baseline
  The brain-PAD score is computed as the difference between estimated brain age and chronological age (brain age minus chronological age).
Complex attention | Baseline
  Attention network test (ANT) is an individually administered computerized task designed to evaluate three attentional components.
Memory and learning | Baseline
  Word list learning test consisting of fifteen semantically non-associated words that is presented consecutively over three trials of immediate recall and a 20-min delayed recall.
Executive function | Baseline
  Executive function is measured by the category verbal fluency test (CVFT).

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Lu, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Tai Po Hospital, Hong Kong, Hong Kong